CLINICAL TRIAL: NCT06238349
Title: Efficacy and Safety of Sunbathing Plus Bifidobacterium for Hyperbilirubinemia in Full-term Neonates: a Prospective Randomized Controlled Study
Brief Title: Hyperbilirubinemia in Full-term Neonates
Acronym: HFN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhuhai Center for Maternal and Child Health Care (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Gaohong Wu, Principal Investigator, Zhuhai Center for Maternal and Child Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GWu; NKRDRC/2022YFC270480 (Other Grant/Funding Number: Yuan Shi)
Record Dates: First submitted 2024-01-23; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Sunbathing; Bifidobacterium; Prevention; Full-term neonates; Hyperbilirubinemia; Randomized controlled trial
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Other): Conventional treatment: Neonates will be placed in an incubator (Ningbo David Medical Device Co., LTD, XHZ model) at 30℃ and relative humidity at 55%. Throughout the study, exclusive breastfeeding and professional care will be provided for the newborns. Newborns requiring phototherapy receive it in the following manner: Phototherapy eye masks (Foshan Forman Medical Technology Co., LTD., Yuesun Mechanical Equipment No. 20160015) and phototherapy diapers (Foshan Baojusheng Medical Equipment Co., LTD., GB/T33280) will be used to cover the eyes and perineum, respectively. Phototherapy was provided via LED blue light continuous irradiation with a wavelength of 425-475nm. All treated neonates will receive continuous phototherapy for 12 hours, then allowe to rest for 6-8 hours, then receive another 12 hours of continuous phototherapy. The decision to continue with further treatment depends on changes in the neonate's jaundice.
  Interventions: Other: Conventional treatment
- Sunbathing group (Experimental): The sunbathing group will receive all interventions prescribed for the control group and assign to sunbathing (placement in a bed next to a sunny window) after birth for one week according to the following plan: Every morning and afternoon neonates will sunbath for 0.5 to 1 hour to avoid excess sun exposure. Healthcare workers will guide and assist families in their preparations. The caregiver will place a black eye patch on the infants to protect the retina, and a cloth will be wrapped around the hands and feet to prevent scratching, but care will be taken that the wrap is not too tight to avoid circulation disorders. Baby boys will have their genitals covered to protect them from sun damage. After feeding, the newborn will be placed on a sunny platform with fully exposed skin and frequent position changes, while the glass of the window prevent injury from UV light exposure.
  Interventions: Other: Sunbathing
- Bifidobacterium group (Experimental): The newborns in the Bifidobacterium group will receive all interventions prescribed for the control group, and also be assigned to orally be given Bifidobacterium triple viable powder (Shanghai Xinyi Pharmaceutical Company, Peifeikang powder, 0.5 g/dose, 3 times/day. Bifidobacterium triple viable powder contains live bacteria of long Bifidobacterium at no less than 1.0 × 107 CFU/g, stored at 2.8℃ away from light) beginning within 24 hours after birth and continuing for 1 week. No sunbathing will be prescribed.
  Interventions: Drug: Oral bifidobacterium triple live powder
- Combination group (Experimental): The combination group will receive all interventions of both the group sunbathing and the Bifidobacterium group as well as all interventions prescribed for the control group.
  Interventions: Other: Sunbathing and the Oral bifidobacterium triple live powder

INTERVENTIONS:
Drug: Oral bifidobacterium triple live powder — The newborns in the Bifidobacterium group will receive all interventions prescribed for the control group, and also were assigned to orally be given Bifidobacterium triple viable powder (Shanghai Xinyi Pharmaceutical Company, Peifeikang powder, 0.5 g/dose, 3 times/day. Bifidobacterium triple viable powder contains live bacteria of long Bifidobacterium at no less than 1.0 × 107 CFU/g, stored at 2.8℃ away from light) beginning within 24 hours after birth and continuing for 1 week. No sunbathing will be prescribed.
  Other Names: Conventional treatment
  Arms: Bifidobacterium group
Other: Sunbathing — The sunbathing group will receive all interventions prescribed for the control group and be assigned to sunbathing (placement in a bed next to a sunny window) after birth for one week according to the following plan: Every morning and afternoon neonates sunbath for 0.5 to 1 hour to avoid excess sun exposure. Healthcare workers will guide and assist families in their preparations. The caregiver will place a black eye patch on the infants to protect the retina, and a cloth will be wrapped around the hands and feet to prevent scratching, but care will be taken that the wrap is not too tight to avoid circulation disorders. Baby boys will have their genitals covered to protect them from sun damage. After feeding, the newborn will be placed on a sunny platform with fully exposed skin and frequent position changes, while the glass of the window prevent injury from UV light exposure.
  Arms: Sunbathing group
Other: Sunbathing and the Oral bifidobacterium triple live powder — The combination group will receive all interventions of both the group sunbathing and the Bifidobacterium group as well as all interventions prescribed for the control group.
  Arms: Combination group
Other: Conventional treatment — Conventional treatment: Neonates will be placed in an incubator (Ningbo David Medical Device Co., LTD, XHZ model) at 30℃ and relative humidity at 55%. Throughout the study, exclusive breastfeeding and professional care will be provided for the newborns. Newborns requiring phototherapy receive it in the following manner: Phototherapy eye masks (Foshan Forman Medical Technology Co., LTD., Yuesun Mechanical Equipment No. 20160015) and phototherapy diapers (Foshan Baojusheng Medical Equipment Co., LTD., GB/T33280) will be used to cover the eyes and perineum, respectively. Phototherapy was provided via LED blue light continuous irradiation with a wavelength of 425-475nm. All treated neonates will receive continuous phototherapy for 12 hours, then allowe to rest for 6-8 hours, then receive another 12 hours of continuous phototherapy. The decision to continue with further treatment depends on changes in the neonate's jaundice.
  Arms: Control group

SUMMARY:
To evaluate the efficacy and safety of sunbathing and Bifidobacterium alone or in combination for full-term neonates with hyperbilirubinemia. The investigators hypothesize that the combination therapy of sunbathing plus Bifidobacterium is safe and effective for prevention and management of hyperbilirubinemia in full-term neonates. The investigators therefore design this prospective, randomized, controlled study to assess the preventive effects of sunbathing combined with Bifidobacterium supplementation on hyperbilirubinemia in full-term neonates. These observations may provide scientific evidence for the use of sunbathing and Bifidobacterium supplementation in the management of hyperbilirubinemia in full-term neonates.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of sunbathing and Bifidobacterium alone or in combination for full-term neonates with hyperbilirubinemia. The investigators hypothesize that the combination therapy of sunbathing plus Bifidobacterium is safe and effective for prevention and management of hyperbilirubinemia in full-term neonates. The investigators therefore design this prospective, randomized, controlled study to assess the preventive effects of sunbathing combined with Bifidobacterium supplementation on hyperbilirubinemia in full-term neonates. A total of 200 neonates treating in Zhuhai Center for Maternal and Child Health Care from Jan. 2024 to Jun. 2024 will be randomized assigned to either trial groups (receiving sunbathing and Bifidobacterium either alone or in combination) or control group receiving traditional therapy. The primary outcome is the incidence of the hyperbilirubinemia and the secondary outcomes include the hospitalization rate, the hospital stays due to hyperbilirubinemia, and the bilirubin levels. Statistical analyses will be performed using ANOVA or chi-square tests, and further pairwise comparisons will be performed using the Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* Term infants with 37 weeks ≤ gestational age < 42 weeks and 2500g ≤ birth weight < 4000g
* Age ≤24 hours
* Stable basic vital signs
* Liver and kidney function normal
* No prior use of antibiotics or ecological agents before specimen collection
* Healthy mothers during pregnancy, with no history of antibiotics or microecological agents before, during, or after childbirth
* Exclusively breastfed
* Informed consent provided voluntarily.

Exclusion Criteria:

* Gestational age <37 weeks or ≥42 weeks
* Complications present with pneumonia, septicemia, or other illness
* Severe immunodeficiency disease present
* Inherited metabolic diseases identified
* Congenital biliary malformations or other organ malformations
* Drug allergies
* History of asphyxiation
* Before enteral feeding, constipation, abdominal distension, diarrhea, vomiting or other gastrointestinal symptoms had appeared
* Enteral feeding was not performed
* Antibiotics or other microecological agents were used
* Isoimmune hemolysis, extravascular hemolysis, polycythemia, erythrocyte enzyme deficiency, erythrocyte morphological abnormality, hemoglobinopathy, etc.
* Hyperbilirubinemia were diagnosed within 24 hours of birth
* Situations that may warrant exclusion as determined by the researcher, such as a guardian with mental illness or frequent changes in living or working environments, which might result in loss of follow-up

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-06-21 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with hyperbilirubinemia | From 1 to 7 days after birth
  Comparisons will be made of the numbers of neonates with hyperbilirubinemia between groups (Sunbathing group vs. Control group, Bifidobacterium group vs. Control group, Combination group vs. Control group, Combination group vs. sunbathing group, Combination group vs. Bifidobacterium group, and Bifidobacterium vs. sunbathing group).

SECONDARY OUTCOMES:
Rate of hospitalization | From 1 to 7 days after birth
  Comparisons will be made in hospitalization rate in the first week of life between groups (sunbathing group vs. Control group, Bifidobacterium group vs. Control group, Combination group vs. Control group, Combination group vs. sunbathing group, Combination group vs. Bifidobacterium group, and Bifidobacterium vs. sunbathing group).
Hospital stays due to hyperbilirubinemia | From 1 to 7 days after birth
  Comparisons will be made in hospital stays due to hyperbilirubinemia in the first week of life between groups (sunbathing group vs. Control group, Bifidobacterium group vs. Control group, Combination group vs. Control group, Combination group vs. sunbathing group, Combination group vs. Bifidobacterium group, and Bifidobacterium vs. sunbathing group).
Participants's bilirubin levels | From 1 to 7 days after birth
  Comparisons will be made in bilirubin levels in the first week of life between groups (sunbathing group vs. Control group, Bifidobacterium group vs. Control group, Combination group vs. Control group, Combination group vs. sunbathing group, Combination group vs. Bifidobacterium group, and Bifidobacterium vs. sunbathing group).

OTHER OUTCOMES:
Numbers of participants with adverse event | From 1 to 7 days after birth
  Neonates in the intervention groups will be monitored for potential side effects, including rash, infection, diarrhea, dehydration, and electrolyte disturbances.
Numbers of participants with single or multiple births | From 1 to 7 days after birth
  Single or multiple births will be collected and compared.
Numbers of participants with intrauterine distress | From 1 to 7 days after birth
  Intrauterine distress will be collected and compared.
Participants's gestational age | From 1 to 7 days after birth
  Gestational age will be collected and compared.
Participants's sex | From 1 to 7 days after birth
  Sex will be collected and compared.
Participants's delivery mode | From 1 to 7 days after birth
  Delivery mode will be collected and compared.
Participants's birth weight | From 1 to 7 days after birth
  Birth weight in kilograms will be collected and compared.
Participants's head circumference | From 1 to 7 days after birth
  Head circumference in centimeter will be collected and compared.
Participants's birth length | From 1 to 7 days after birth
  Birth length in centimeter will be collected and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, M.D., Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Zhuhai Center for Maternal and Child Health Care, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
We want to share IPD after we've done our research.